CLINICAL TRIAL: NCT02540928
Title: A Cancer Research UK Randomised, Double Blind, Placebo Controlled Phase IIa Trial of AMG 319 Given Orally as a Neoadjuvant Therapy in Patients With Human Papillomavirus (HPV) Positive and Negative Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: AMG 319 in HPV Positive and Negative HNSCC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety Reasons
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRUKD/15/004
Record Dates: First submitted 2015-08-25; First posted 2015-09-04 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Human Papillomavirus (HPV); Positive or Negative Head and Neck Squamous Cell Carcinoma (HNSCC) of the Hypopharynx, Oropharynx, Oral Cavity, Supraglottis or Larynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AMG 319 Hydrate (Experimental): Up to 36 patients will be randomised into the Active Treatment arm to receive AMG 319 400 mg once daily administered orally for a minimum of 20 days and a maximum of 29 days prior to resection surgery
  Interventions: Drug: AMG 319 hydrate
- Placebo (Placebo Comparator): Up to 18 patients will be randomised into the Placebo arm to receive Placebo once daily administered orally for a minimum of 20 days and a maximum of 29 days prior to resection surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AMG 319 hydrate
  Arms: AMG 319 Hydrate
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether a drug called AMG 319 has an effect on a patient's own immune response to head and neck cancer squamous cell carcinoma (HNSCC). This study is specifically for patients who are having surgery to treat their HNSCC

DETAILED DESCRIPTION:
Cancers use 'defence mechanisms' to hide from the immune system and teach the immune system not to destroy cancer cells. AMG 319 works by blocking these defence mechanisms in the tumour. It targets and blocks an important protein called PI3K delta.

In the laboratory this leads to removal of a group of inhibitory immune cells. Releasing the immune brakes leads to immune attack and destruction of cancer cells.

AMG 319 looks promising in laboratory studies and in a very early study in a small number of patients with leukaemia and we now wish to find out if it will be useful in treating patients with head and neck cancer.

This study is a randomised, doubleblind, placebo controlled Phase II trial looking at the effects of giving AMG 319 to patients with either human papilloma virus (HPV) positive or negative head and neck cancer squamous cell carcinoma (HNSCC). We propose to treat patients prior to resection surgery so that we can study the effect of AMG 319 on the cancer in fine detail.

Approximately 54 patients with HPV positive or negative HNSCC of the hypopharynx, oropharynx, oral cavity, supraglottis or larynx will be entered into the study. Patients will be randomly assigned to one of two treatment groups and will receive between 20 and 29 days of oral dosing with AMG 319 or placebo immediately before resection surgery.

ELIGIBILITY:
Inclusion criteria:

1. Histologically proven HNSCC of the hypopharynx, oropharynx, oral cavity, supraglottis or larynx (except T1 glottic tumours) for whom surgery with curative intent ± post operative radiotherapy or chemoradiotherapy is considered the primary treatment of choice. Surgery should be scheduled to take place no sooner than 21 days and no later than 30 days post first dose of AMG 319 or placebo.

   Patients presenting with recurrence can be considered for inclusion, as long as their previous treatment did not include radiotherapy ± chemotherapy or any other anti cancer therapy i.e. treated with surgery alone and this did not take place within 6 months prior to trial entry.

   Patients presenting with a second primary HNSCC can be considered for inclusion, as long as any previous radiotherapy, chemotherapy or any other anti cancer therapy was completed more than 5 years prior to trial entry.
2. Patients considered fit to undergo curative resection surgery.
3. Haematological and biochemical indices within the ranges shown below:

   Laboratory Test Value required

   Haemoglobin (Hb) ≥100 g/L

   Absolute neutrophil count ≥1.5 x 109/L

   Platelet count ≥100 x 109/L

   Bilirubin ≤1.5 x upper limit of normal (ULN) Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 x ULN

   Alkaline Phosphatase (alk phos/ALP) ≤2.5 x ULN

   Amylase ≤2.0 x ULN

   Calculated creatinine clearance (using the Wright or Cockcroft-Gault formula) ≥50 mL/min
4. 18 years or over at the time informed consent is given.
5. Written (signed and dated) informed consent and capable of co-operating with treatment and follow up.

Exclusion criteria:

1. Prior radiotherapy, immunotherapy, chemotherapy or other anti-cancer therapy (excluding surgery) for current HNSCC.
2. Patients should be excluded from the trial if they have active or previous malignancies of other types which in the Investigator's opinion would mean they are not a good candidate for the clinical trial.
3. Female patients who are able to become pregnant (or already pregnant or lactating). However, those patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral; injected or implanted hormonal contraception and condom; have an intra uterine device and condom; diaphragm with spermicidal gel and condom) effective at the first administration of AMG 319, throughout the trial and for 6 months afterwards are considered eligible.
4. Male patients with partners of child bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] effective at the first administration of AMG 319, throughout the trial and for 6 months afterwards). Men with pregnant or lactating partners must be advised to use barrier method contraception (for example: condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
5. Patients unable to swallow oral medications (trial medication must not be chewed, crushed, dissolved or divided).
6. Major thoracic or abdominal surgery from which the patient has not yet recovered.
7. At high medical risk because of non malignant systemic disease including active uncontrolled infection.
8. Active or uncontrolled auto immune disease which may require systemic immunomodulator therapy during the trial treatment period. Exceptions to this are atopic dermatitis and psoriasis not requiring systemic treatment.
9. Long term use of systemic corticosteroids with the exception of replacement treatment. Discontinuation of steroid use within seven days prior to receiving the first dose of AMG 319 or placebo would be acceptable. Inhaled and topical steroids are permitted.
10. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV). If there is clinical suspicion of infection this must be ruled out by appropriate serological and PCR testing.
11. QTc >470 msec (Friderica [QTc F] correction) or a history or family history of QT prolongation.
12. Regular and/or prolonged treatment with medications known to cause QTc interval prolongation within seven days prior to receiving the first dose of AMG 319 or placebo.
13. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase IIa trial of AMG 319. Participation in an observational trial or interventional clinical trial which does not involve administration of an IMP would be acceptable.
14. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-10; Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

PRIMARY OUTCOMES:
Changes in CD8+ effector T cell numbers in tumour tissue | Screening and Surgery
Treatment emergent adverse events | Assessed until 60 days after a patients last dose

SECONDARY OUTCOMES:
Steady State AMG 319 concentration in blood | Days 8, 15 pre dose & Day 22
Changes in tumour size | Screening and Pre-surgery

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Aintree University Hospital - Clatterbridge Cancer Centre, Liverpool
  - Churchill Hospital, Blenheim H&N Unit, Oxford
  - Poole Hospital, Poole
  - Queen Alexandra Hospital, Department of Oral and Maxillofacial Surgery, Portsmouth
  - Southampton General Hospital, Southampton